CLINICAL TRIAL: NCT04085549
Title: Effects of a Berry Oil Cream on Atopic Eczema and Skin
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was ceased due to Covid-19 epidemia.
Sponsor: Petra Larmo (Industry)
Collaborators: Cliniscan Ltd (Unknown)
Responsible Party: Sponsor-Investigator, Petra Larmo, Ph.D., R&D Manager, Aromtech Ltd.
Organization: Aromtech Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BOAE
Record Dates: First submitted 2019-09-09; First posted 2019-09-11 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2021-01

CONDITIONS: Atopic Dermatitis Eczema

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Study has two parts. In part 1 the participants, care provider and outcome assessor know which treatment is given to each skin area. In part 2 participant, care provider, investigator and outcome assessor do not know which treatment is given to each skin area. Masking is done by identical cream tubes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Berry Oil Cream (Experimental): Study part 1: Administered to a chosen eczema lesion on randomized body half 1-2 times/d or more frequently (use reported to study logbook) for two weeks. Also administered to forearm (randomized body half) twice/d for two weeks. Study part 2: Administered to randomized body half 1-2 times/d for five weeks.
  Interventions: Device: Berry Oil Cream
- Control (No Intervention): Study part 1: A chosen eczema lesion on randomized body half is an untreated control for two weeks. Also one forearm (on randomized body half) is a control with no treatment for two weeks.
- Reference cream (Active Comparator): A commercial reference cream, not containing berry and plant oils. Study part 2: Administered to randomized body half 1-2 times/d for five weeks.
  Interventions: Other: Reference Cream

INTERVENTIONS:
Device: Berry Oil Cream — Cream containing berry and plant oils and humectants; a medical device product in development
  Arms: Berry Oil Cream
Other: Reference Cream — Commercial refence cream not containing berry and plant oils.
  Arms: Reference cream

SUMMARY:
Atopic eczema is a chronic inflammatory skin disease associated with itch and inflammatory lesions in typical skin areas. The objective of this study is to investigate the effects of a cream containing berry and plant oils and humectants on atopic eczema and dry skin.

ELIGIBILITY:
Inclusion Criteria:

* Atopic Eczema (mild or medium severity)

Exclusion Criteria:

* Other serious skin conditions (for example psoriasis)
* Known hypersensitivity to ingredients of the study creams
* Medication seriously affecting immune function

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2019-10-09 (Actual); Primary Completion 2020-04-15 (Actual); Study Completion 2020-04-15 (Actual)

PRIMARY OUTCOMES:
Change in severity of atopic eczema | Part 1: Baseline, 2 weeks. Part 2: Baseline, 5 weeks
  Objective local Scoring Atopic Dermatitis (SCORAD) index. Scale range for objective local scorad in study part 1 (chosen eczema lesion) 0-63, in study part 2 (body half) 0-73. Decrease indicates better outcome/ milder symptoms.
Change in severity of symptoms | Part 1: Baseline, 2 weeks. Part 2: Baseline, 2 weeks, 5 weeks
  Modified Patient Oriented Eczema Measure (POEM) questionnaire. Scale range: 0-24. Decrease indicates better outcome/ milder symptoms.
Change in sensation of itch | Part 1: Baseline, 2 weeks. Part 2: Baseline, 2 weeks, 5 weeks
  Visual Analog Scale (VAS) evaluation. Scale range 0-10. Decrease indicates better outcome/ milder symptoms.
Change in transepidermal water loss (TEWL) | Part 1: Baseline, 2 weeks. Part 2: Baseline, 2 weeks, 5 weeks
  Measurement of TEWL (g/m2h)
Change in skin hydration | Part 1: Baseline, 2 weeks. Part 2: Baseline, 2 weeks, 5 weeks
  Measurement of moisture (capacitance, proportional to water content of skin)
Change in skin pH | Part 1: Baseline, 2 weeks. Part 2: Baseline, 2 weeks, 5 weeks
  Measurement of skin pH

SECONDARY OUTCOMES:
Change in symptoms of itching, dryness, flaking of skin | Part 1: Baseline, 2 weeks. Part 2: Baseline, 2 weeks, 5 weeks
  Symptom logbooks: daily scoring from 0 (no symptoms) to 3 (severe symptoms)

CONTACTS AND LOCATIONS:
Overall Officials: Risto Oksman, MD, Principal Investigator — Cliniscan Ltd
Locations (1):
- Mehiläinen (Private Clinic), Turku, Finland

IPD SHARING:
Plan to Share IPD: No